CLINICAL TRIAL: NCT07052604
Title: Antibiotic Treatment for Pneumonia Caused by Stenotrophomonas Maltophilia in ICU Patients
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0055_STENO
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Pneumonia, Ventilator-Associated; Stenotrophomonas Maltophilia; Intensive Care Units; Anti-Bacterial Agents; Drug Resistance, Bacterial
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study looks at how different antibiotic treatments affect patients in intensive care who have pneumonia caused by the bacteria Stenotrophomonas maltophilia. It compares using one antibiotic versus two antibiotics, and treatment lengths of 7 days versus 14 days, to see which approach helps patients survive better. The study also examines how resistant the bacteria are to antibiotics and how often the pneumonia comes back.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years)
* Hospitalized in Medical Intensive Care Unit between January 1, 2018, and December 31, 2023
* Intubated and mechanically ventilated
* Diagnosed with ventilator-associated pneumonia caused by Stenotrophomonas maltophilia

Exclusion Criteria:

* Patients under 18 years old
* Patients who refuse the use of their data for research purposes

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients admitted to the Medical Intensive Care Unit (ICU) between January 2018 and December 2023 who are intubated and mechanically ventilated, and who develop ventilator-associated pneumonia caused by Stenotrophomonas maltophilia. These patients represent a critical care group at high risk for serious infections with multidrug-resistant bacteria.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
patient survival based on the antibiotic treatment strategy used (monotherapy vs. combination therapy and 7 vs. 14 days duration). | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Saint-Denis, Saint-Denis, France, France